CLINICAL TRIAL: NCT05645913
Title: Association of Obesity and Cardiovascular Outcomes in Patients With Atrial Fibrillation : a Korean Nationwide Cohort Study
Brief Title: Association of Obesity and Cardiovascular Outcomes in Atrial Fibrillation
Acronym: Paradox
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Kwang-No Lee, Professor, Ajou University School of Medicine
Other Study IDs: AJOUIRB-EXP-2021-398
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation; Obesity; Prognosis; Anticoagulants
MeSH Terms: conditions — Atrial Fibrillation; Obesity | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial fibrillation with oral anticoagulant: patients who were newly receiving an oral anticoagulant for atrial fibrillation during study period
  Interventions: Drug: Oral anticoagulant

INTERVENTIONS:
Drug: Oral anticoagulant — Oral anticoagulant that was continued at least 25days, inculding warfarin and new oral anticoagulant (NOAC)
  Other Names: Oral anticoagulant medication

SUMMARY:
In this study, the investigators evaluated the association between various measures of adiposity [BMI and waist circumference (WC)] and clinical outcomes in Asian patients with AF who were prescribed OAC, using a nationwide population based cohort.

DETAILED DESCRIPTION:
This retrospective nationwide cohort study used administrative claims data from the Korean National Health Insurance Service (NHIS) and the combined health check-up database of the National Health Insurance Corporation between 2013 and 2020.

The investigators included oral anticoagulant (OAC) new users diagnosed with atrial fibrillation (AF) between January 2015 and December 2020. Patients aged <20 years, those who were regarded as valvular AF patients (patients with mitral stenosis or prosthetic heart valve), those with possible alternative indications for OAC (pulmonary embolism, deep vein thrombosis, or recent joint replacement surgery), and those with cancer were excluded from the analysis.

The follow-up period was defined as the time from the index date (date of OAC prescription) to each outcome event, date of death, or end of the study period (December 31, 2020), whichever came first.

Patients' demographic data, comorbidities, concomitant medications, and income level were collected from the Korean NHIS database. The recent health check-up data from the index date was also ascertained, including height, weight, waist circumference, blood pressure, health surveys, and laboratory exam. Health survey included family history, smoking history, alcohol history, and the level of individual physical activity. The investigators defined the proportion of medical use by calculating formula with the recuperation cost and the number of the visit to hospitals.

According to BMI following the World Health Organization recommendation for Asian population, study patients were categorized into 5 groups: underweight, <18.5 kg/m2; normal range, 18.5 to <23 kg/m2; overweight, 23 to <25 kg/m2; obese I, 25 to <30 kg/m2; and obese II, ≥30 kg/m2[4].

During the follow-up period, the investigators assessed 3 clinical outcomes, including thromboembolism, major bleeding, all-cause death, and a composite clinical outcome of thromboembolism+major bleeding+all-cause death. Major bleeding included the brain hemorrhage and gastrointestinal bleeding. Clinical outcomes were mainly defined by the the International Classification of Diseases, 10th revision (ICD-10). Patients were censored at the clinical outcomes, the discontinuation of index OAC treatment, or the end of the study period (December 31, 2020), whichever came first.

Continuous variables are presented as mean±SD or median (interquartile ranges). Categorical variables are presented as numbers and percentages. Baseline characteristics were compared across 5 BMI categories with a linear trend test using a generalized linear model for continuous variables and the Cochran-Armitage trend test for categorical variables. The incidence rates of clinical outcomes were calculated based on the number of events during the follow-up period divided by 100 person-years at risk.

For the primary analyses to evaluate the association between BMI and clinical outcomes in AF patients treated with OAC, the investigators conducted 2 types of analyses: (1) BMI as a continuous variable and (2) BMI as a categorical variable by predefined BMI ranges. First, the association between BMI as a continuous variable (per 5 kg/m2 increase) and clinical outcomes was evaluated using a Cox proportional hazard model to derive unadjusted and adjusted hazard ratios (HRs). Adjusted cubic spline curves were used to visualize the relationship between BMI and the risk of clinical outcomes. Second, the association between different BMI categories and clinical outcomes was explored using adjusted Cox proportional hazard models. Patients with a normal range of BMI defined as 23 to <25 kg/m2 were used as the reference group. Covariates in the multivariable analysis included age, sex, CHA2DS2-VASc score, comorbidities, renal function, use of antiplatelet agents, and OAC treatment (warfarin or non-vitamin K antagonist OAC [NOAC]).

All analyses were 2 tailed, and P<0.05 was considered significant. Statistical analyses were conducted with R-statistics.

ELIGIBILITY:
Inclusion Criteria:

* Oral anticoagulant (OAC) new users diagnosed with atrial fibrillation (AF) between January 2015 and December 2020

Exclusion Criteria:

* Patients aged <20 years
* Valvular AF patients
* Possible alternative indications for OAC (pulmonary embolism, deep vein thrombosis, or recent joint replacement surgery)
* Cancer patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This retrospective nationwide cohort study used administrative claims data from the Korean National Health Insurance Service (NHIS) and the combined health check-up database of the National Health Insurance Corporation between 2013 and 2020.
  We included oral anticoagulant (OAC) new users diagnosed with atrial fibrillation (AF) between January 2015 and December 2020. Patients aged <20 years, those who were regarded as valvular AF patients (patients with mitral stenosis or prosthetic heart valve), those with possible alternative indications for OAC (pulmonary embolism, deep vein thrombosis, or recent joint replacement surgery), and those with cancer were excluded from the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 56272 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of Outcomes | 5 years
  Thromboembolism+Bleeding+Death

SECONDARY OUTCOMES:
Thromboembolism | 5 years
  Stroke, Myocardial infarction
Bleeding | 5 years
  Intracranial hemorrhage, Hospitalization for GI bleeding
Death | 5 years
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-No LEE, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim MS, Kim WJ, Khera AV, Kim JY, Yon DK, Lee SW, Shin JI, Won HH. Association between adiposity and cardiovascular outcomes: an umbrella review and meta-analysis of observational and Mendelian randomization studies. Eur Heart J. 2021 Sep 7;42(34):3388-3403. doi: 10.1093/eurheartj/ehab454. PMID 34333589
- [Result] Lee SR, Choi EK, Jung JH, Park SH, Han KD, Oh S, Lip GYH. Body Mass Index and Clinical Outcomes in Asian Patients With Atrial Fibrillation Receiving Oral Anticoagulation. Stroke. 2021 Jan;52(2):521-530. doi: 10.1161/STROKEAHA.120.030356. Epub 2021 Jan 11. PMID 33423512
- [Result] Park SJ, Ha KH, Kim DJ. Body mass index and cardiovascular outcomes in patients with acute coronary syndrome by diabetes status: the obesity paradox in a Korean national cohort study. Cardiovasc Diabetol. 2020 Nov 10;19(1):191. doi: 10.1186/s12933-020-01170-w. PMID 33172464